CLINICAL TRIAL: NCT00357045
Title: Antidepressant Prophylaxis for Interferon-Induced Depression: Efficacy of Paroxetine; THE HEPDEP II STUDY
Brief Title: Antidepressant Prophylaxis for Interferon-Induced Depression: Efficacy of Paroxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 05-1002
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2003-12

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
Objectives:

1. To determine whether paroxetine can prevent major depression in patients with hepatitis C (HCV) who are receiving pegylated-interferon (Peg-IFN).
2. To determine whether paroxetine can prevent subsyndromal increases in depression and anxiety in patients with HCV who are receiving Peg-IFN.
3. To determine whether paroxetine can prevent a significant change in the health related quality of life in patients with HCV who are receiving Peg-IFN.
4. To determine whether paroxetine improves compliance with Peg-IFN therapy for HCV.
5. To determine whether paroxetine enables patients to complete Peg-IFN therapy for HCV who might otherwise require a dose reduction or discontinuation because of neuropsychiatric side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* diagnosis of hepatitis C
* agree to participate in the study with written informed consent
* plan to undergo treatment with Peg-IFN + Ribavirin
* compensated liver disease (hemoglobin value > 12 gm/dL for females or > 13 gm/dL for males, WBC > 3000/mm3, platelets > 70,000/mm3, albumin > 3.0 g/dL or within 20% of LLN, Serum creatinine < 1.4 mg/dL, thyroid stimulating hormone within normal limits
* confirmation from female patients that adequate contraception is being practiced during treatment period and for 6 months after discontinuation of therapy
* confirmation from male patients that acceptable contraception is being practiced

Exclusion Criteria:

* hypersensitivity to IFN, RBV, or paroxetine
* chronic liver disease other than chronic HCV
* hemolytic anemia from any cause including hemoglobinopathies
* evidence of advance liver disease
* any preexisting medical condition that could interfere with participation in the protocol
* evidence of cardiac ischemia, a significant unstable cardiac arrhythmia, heart failure, recent coronary artery surgery, uncontrolled HTN, unstable angina, or MI within past 12 months
* clinically significant retinal abnormalities
* substance abuse (must have abstained from abusing substance for at least 6 months)
* diagnosis of major depression in the past 6 weeks
* currently receiving full therapeutic dose of antidepressant medications
* diagnosis of bipolar disorder
* active psychotic condition
* active delirium
* pregnant female patients, men whose sexual partner is currently pregnant, and men and women who are not practicing adequate contraception
* female patients who are actively breast feeding
* patients with a known history of non-compliance with medical treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: J. K. Moles, M.D., Principal Investigator — Salem VA Medical Center